CLINICAL TRIAL: NCT05989828
Title: Phase Ib Clinical Trial of Autologous Anti-NY-ESO-1 TCR-Engineered T Cells in Patients With Relapsed/Refractory Locally Advanced or Metastatic NY-ESO-1-Expressing Triple Negative Breast Cancer
Brief Title: A2-ESO-1 TCR-Engineered T Cells for Relapsed/Refractory Advanced or Metastatic NY-ESO-1 Overexpression Positive Triple Negative Breast Cancer
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Pending Protocol Amendment Approval
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1B-23-1; NCI-2023-04697 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1B-23-1 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2023-06-27; First posted 2023-08-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — aldesleukin; Biopsy; Specimen Handling; Cyclophosphamide; fludarabine; Leukapheresis; Magnetic Resonance Spectroscopy; High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (A2-ESO-1 TCR-T cells) (Experimental): Patients undergo leukapheresis on day -28 then receive cyclophosphamide IV over 1 hour on days -7 and -6 followed by fludarabine IV over 30 minutes on days -5 to -1. Patients then receive A2-ESO-1 TCR-T cells IV over 30 minutes on day 0 followed by aldesleukin IV over 15 minutes on days 0 to 2. Patients also undergo blood sample collection and CT scans throughout the study. Additionally, patients may undergo a breast biopsy, a mammogram, breast MRI, and breast US at screening and follow up, and ECHO or MUGA at screening.
  Interventions: Biological: Aldesleukin; Biological: Anti-HLA-A2/NY-ESO-1 TCR-transduced Autologous T Lymphocytes; Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Cyclophosphamide; Procedure: Echocardiography; Drug: Fludarabine; Procedure: Leukapheresis; Procedure: Magnetic Resonance Imaging; Procedure: Mammogram; Procedure: Multigated Acquisition Scan; Procedure: Ultrasound Imaging

INTERVENTIONS:
Biological: Aldesleukin — Given IV
  Other Names: 125-L-Serine-2-133-interleukin 2; Proleukin; r-serHuIL-2; Recombinant Human IL-2; Recombinant Human Interleukin-2
Biological: Anti-HLA-A2/NY-ESO-1 TCR-transduced Autologous T Lymphocytes — Given IV
  Other Names: Anti-HLA-A2/NY-ESO1 TCR-transduced Autologous T cells; Autologous Anti-HLA-A2/NY-ESO1 TCR-transduced T Lymphocytes; Autologous HLA-A2/NY-ESO-1-specific TCR Gene-transduced T-lymphocytes
Procedure: Biopsy — Undergo biopsy of breast tumor
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Procedure: Echocardiography — Undergo ECHO
  Other Names: EC
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Procedure: Leukapheresis — Undergo leukapheresis
  Other Names: Leukocytopheresis; Therapeutic Leukopheresis
Procedure: Magnetic Resonance Imaging — Undergo breast MRI
  Other Names: Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: Mammogram — Undergo mammogram
Procedure: Multigated Acquisition Scan — Undergo MUGA scan
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Procedure: Ultrasound Imaging — Undergo ultrasound of breast
  Other Names: 2-Dimensional Grayscale Ultrasound Imaging; 2-Dimensional Ultrasound Imaging; 2D-US; Ultrasonography; Ultrasound; Ultrasound Test; Ultrasound, Medical; US

SUMMARY:
This phase Ib trial tests the safety, side effects and best dose of anti-HLA-A2/NY-ESO-1 T-cell receptor (TCR)-transduced autologous T lymphocytes (A2-ESO-1 TCR-T cells) in treating patients with NY-ESO-1 overexpression positive triple negative breast cancer (TNBC) that has come back after a period of improvement (relapsed/recurrent) or that does not respond to treatment (refractory), and that may have spread from where it first started (primary site) to nearby tissue, lymph nodes (advanced) or to other places in the body (metastatic). NY-ESO-1 is an antigen found on the surface of many different types of tumor cells including TNBC. Antigens make it possible for immune cells to recognize and kill germ cells that invade the body, however, it is more difficult for immune cells to recognize antigens on tumor cells. T cells are a special type of immune cell in the blood. These T cells may be trained to recognize the NY-ESO-1 antigen on tumor cells, allowing the T cells to attack and kill those tumor cells. The A2-ESO-1 TCR-T cells are T cells that have been removed from the patient's blood through a process called leukapheresis and then changed in the laboratory to recognize NY-ESO-1 on tumor cells. When given back to the patient, these A2-ESO-1 TCR-T cells find and attack tumor cells that express NY-ESO-1. Chemotherapy drugs, such as cyclophosphamide and fludarabine, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. They are given before the T cells to support optimum activity of the A2-ESO-1 TCR-T cells. IL-2 (aldesleukin) is in a class of drugs known as cytokines. It is a man-made version of a naturally occurring protein that stimulates the body to produce other chemicals which increase the body's ability to fight cancer. A2-ESO-1 TCR-T cells may kill more tumor cells in patients with recurrent or refractory advanced or metastatic TNBC that overexpresses NY-ESO-1.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of anti-HLA-A2/NY-ESO-1 TCR-transduced autologous T lymphocytes (A2-ESO-1 TCR-engineered T cells) in patients with relapsed/refractory locally advanced or metastatic TNBC that overexpresses NY-ESO-1 by using the Bayesian optimal interval (BOIN) design.

II. To determine the dose-limiting toxicities (DLTs) of A2-ESO-1 TCR-engineered T cells in patients with relapsed/refractory locally advanced or metastatic TNBC that overexpresses NY-ESO-1, as assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version (v)5.0.

SECONDARY OBJECTIVES:

I. To evaluate the antitumor activity of A2-ESO-1 TCR-engineered T cells, as assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.

II. To evaluate the immunological activity (i.e., persistence, function) of A2-ESO-1 TCR-engineered T cells.

EXPLORATORY OBJECTIVE:

I. To evaluate the correlative markers of A2-ESO-1 TCR-engineered T cells, including but not limited to PD-L1 expression and immune cell populations such as regulatory T cells (Tregs) and tumor-associated macrophages (TAMs).

OUTLINE: This is a dose-escalation study of A2-ESO-1 TCR-T cells.

Patients undergo leukapheresis on day -28 then receive cyclophosphamide intravenously (IV) over 1 hour on days -7 and -6 followed by fludarabine IV over 30 minutes on days -5 to -1. Patients then receive A2-ESO-1 TCR-T cells IV over 30 minutes on day 0 followed by aldesleukin IV over 15 minutes on days 0 to 2. Patients also undergo blood sample collection and computed tomography (CT) scans throughout the study. Additionally, patients may undergo a breast biopsy, a mammogram, breast magnetic resonance imaging (MRI), and breast ultrasound (US) at screening and follow up, and echocardiography (ECHO) or multi-gated acquisition scan (MUGA) at screening.

After completion of study treatment, patients are followed up at 3, 6, and 12 months and then yearly for up to 15 years or until disease progression, voluntary study withdrawal or study discontinuation, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Female aged >= 18 years
* Histologically confirmed advanced or metastatic TNBC that have relapsed on or are refractory to 2 or more lines of standard-of-care therapy including immune checkpoint inhibitors, chemotherapy, trastuzumab deruxtecan (TDX-d) and poly-ADP ribose polymerase (PARP) inhibitors if indicated, but less than 4 lines of total therapies. TNBC is defined as estrogen receptor (ER) and progesterone receptor negative (< 10% immunohistochemistry [IHC] staining) and HER2 negative (IHC 1+ or 0 AND/OR in situ hybridization negative based on:

  * Single-probe average HER2 copy number < 4.0 signals/cell
  * Dual-probe HER2/CEP17 ratio < 2.0 with an average HER2 copy number < 4.0 signals/cell)
* HLA-A2+ and tumoral overexpression of NY-ESO-1 (2 to 3+ IHC staining in > 50% of cells)
* Have measurable disease based on RECIST 1.1
* Life expectancy >= 6 months
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Hemoglobin >= 9.0 g/dL (transfusions permitted)
* Absolute neutrophil count (ANC) >= 1500/mm^3
* Platelet count >= 100,000/mm^3
* Creatinine (Cr) < 2 x upper limit of normal (ULN), and Cr clearance (CrCl) >= 50 mL/min by Cockcroft and Gault
* Alanine transaminase (ALT) and aspartate transaminase (AST) < 2 x ULN (Patients with liver metastases whose ALT/AST are < 5 x ULN are eligible for enrollment)
* Bilirubin < 2 x ULN
* White blood cell (WBC) count > 2500/uL and < 15000/uL
* Lymphocyte count >= 500/uL
* Cardiac ejection fraction >= 50%
* Negative serum pregnancy (human chorionic gonadotropin [beta-hCG]) test within 7 days of leukapheresis for women of childbearing potential (WOCBP). WOCBP must be willing to use a highly effective method of contraception for the course of the study through 90 days after A2-ESO-1 TCR-engineered T cell infusion
* Willing and able to provide written informed consent for the study
* Willing to provide biopsy tissues and blood samples as required by the study

Exclusion Criteria:

* Radiation therapy, chemotherapy, or non-cytotoxic investigational agent within 2 weeks of leukapheresis
* Received cyclophosphamide within the past 4 months
* Evidence of New York Heart Association class III or greater cardiac disease
* History of myocardial infarction, stroke, ventricular arrhythmia, or symptomatic conduction abnormality within the past 12 months
* History of congenital QT prolongation
* Absolute QT interval of > 470 msec in the presence of > 4.0 mEq/L potassium and > 1.8 mg/dL magnesium
* Brain or leptomeningeal metastases
* Females who are pregnant or breastfeeding
* Hypersensitivity or intolerance to cyclophosphamide, fludarabine, or their components
* Alcoholic liver disease or other hepatic disease with the exception of liver metastases
* History of gastrointestinal bleeding, ulceration, or perforation
* Any severe and/or uncontrolled medical conditions or other conditions that could affect participation in the study, such as severely impaired lung function, any active (acute or chronic) or uncontrolled infection/disorders, and non-malignant medical illnesses that are uncontrolled or whose control may be jeopardized by the study treatment
* Current use of medications that interact with or compromise the immune system such as steroid doses > 10 mg/day prednisone or equivalent daily within 2 weeks before leukapheresis
* History of immunodeficiency disease or autoimmune disease, with exceptions such as Hashimoto's thyroiditis / hypothyroidism, or controlled Type 1 diabetes
* Have any active and uncontrolled infection.
* Active hepatitis B or hepatitis C infection or seropositive for hepatitis B, and hepatitis C antibody unless antigen negative. If hepatitis C antibody test is positive, then patients must be tested for the presence of antigen by RT-PCR and be HCV RNA negative
* Human immunodeficiency virus (HIV) infection or seropositive for HIV antigens
* Concurrent use of any complementary or alternative medicines
* Unwilling or unable to comply with the study protocol
* Prior major surgery that requires general anesthesia must be completed at least 4 weeks before leukapheresis and surgery that requires local anesthesia (except for study tissue sample collection) must be completed at least 2 weeks before leukapheresis and surgery that requires local anesthesia (except for study tissue sample collection) must be completed at least 2 weeks before leukapheresis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12-17 (Actual); Primary Completion 2026-12-17 (Estimated); Study Completion 2027-12-17 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of anti-HLA-A2/NY-ESO-1 T-cell receptor (TCR)-transduced autologous T lymphocytes (A2-ESO-1 TCR-engineered T cells) | Up to 8 weeks after A2-ESO-1 TCR-engineered T cell infusion
  Will employ the Bayesian optimal interval to find the MTD.
Incidence of dose-limiting toxicities | Up to 8 weeks after A2 ESO-1 TCR-engineered T cell infusion
  Defined as any treatment-related death or any greater than or equal to grade 3 adverse event (AE) as assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0.

SECONDARY OUTCOMES:
Antitumor activity | At pre-treatment and 6 months post-treatment
  Antitumor activity will be assessed by RECIST 1.1. Complete Response (CR) = disappearance of all target lesions, Partial Response (PR) = at least a 30% decrease in the sum of the longest diameter of target lesions, using the baseline sum longest diameter as a reference, Stable Disease (SD) = Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for Progressive Disease (PD) using the smallest sum longest diameter since treatment start as reference, PD = At least a ≥20% increase in the sum of the longest dimensions of the target lesions taking as a reference the smallest sum of the longest dimensions recorded since the treatment started, or the appearance of one or more new lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Change in PD-1 expression on T cells | At pre-treatment and 6 months post-treatment
  Levels of PD-1 expression on T cells will be monitored. Post-treatment biomarker measurements will be compared to the pre-treatment values using a one-sided paired t-test and nonparametric Wilcoxon signed-rank test.
Change in NY-ESO-1-specific TCR-engineered T cells | At pre-treatment and 6 months post-treatment
  Levels of NY-ESO-1-specific TCR-engineered T cells will be monitored to determine whether these T cells are persistent. Post-treatment biomarker measurements will be compared to the pre-treatment values using a one-sided paired t-test and nonparametric Wilcoxon signed-rank test.
Change in regulatory T cells (Treg) | At pre-treatment and 6 months post-treatment
  Because NY-ESO-1-specific TCR-engineered CD4+ T cells may differentiate into Treg cells, levels of Treg cells will be monitored. Post-treatment biomarker measurements will be compared to the pre-treatment values using a one-sided paired t-test and nonparametric Wilcoxon signed-rank test.

CONTACTS AND LOCATIONS:
Overall Officials: Daphne Stewart, MD, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States